CLINICAL TRIAL: NCT02106780
Title: An Open Label Study to Evaluate the Pharmacokinetics of ASP1707 After a Single Oral Dose of 14C-labeled ASP1707 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Effect of ASP1707 on the Bodies of Healthy Male Subjects After a Single Dose of Radioactive ASP1707
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1707-CL-0021; 2011-001701-27 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Pharmacokinetics of ASP1707
Keywords: Phase 1; Healthy subjects; Excretion; 14C-labeled ASP1707

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: ASP1707 (Experimental)
  Interventions: Drug: 14C-labeled ASP1707

INTERVENTIONS:
Drug: 14C-labeled ASP1707 — oral

SUMMARY:
Subjects receive a single oral dose of radioactive ASP1707 on Day 1. Blood, plasma, urine and feces samples are collected for analysis of 14C-radioactivity and ASP1707. Metabolites are collected until at least 144 hours after dosing.

DETAILED DESCRIPTION:
Subjects are admitted to the clinic on Day -1 and receive a single oral dose of 14C-labeled ASP1707 on Day 1. They remain in the clinic for 6 days and are discharged on Day 7 if sufficient recovery of administered radioactivity is achieved, or the total excretion (urine + feces) per 24 hours is less than 1% of the administered dose during 2 consecutive 24-hour intervals. If these conditions are not met, the residential period may be prolonged for a maximum of 3 days. If after this time one of the conditions is still not met, subjects are requested to continue collecting their urine and/or feces at home for another 2 days. If after these additional 2 days one of the conditions is still not met, the condition of recovery of radioactivity is disregarded. Therefore only the total excretion condition is to be met by collecting 24-hour intervals for urine and feces once a week for up to 2 weeks. If the excretion condition is still not met after this time, no further samples are collected and the subject is discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be surgically sterilized and use condoms or must practice an effective contraceptive method to prevent pregnancies.
* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2.
* Regular defecation pattern (minimum once per day).

Exclusion Criteria:

* Any of the liver function tests above the upper limit of normal.
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a clinical study in the previous year.
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit.
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit.
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit.
* Positive serology test for Hepatitis B Surface Antigen (HBsAg), anti Hepatitis A Virus (HAV) Immunoglobulin M (IgM), anti Hepatitis C Virus (HCV) or anti Human Immunodeficiency Virus (HIV) 1+2.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Radioactivity in whole blood measured by Area under the plasma concentration - to time = infinity (AUCinf) | Day -1 until at least Day 7
Radioactivity in whole blood measured by Area under the plasma concentration - time curve to the last quantifiable concentration (AUClast) | Day -1 until at least Day 7
Radioactivity in whole blood measured by Maximum concentration (Cmax) | Day -1 until at least Day 7
Radioactivity in whole blood measured by Time to Attain Cmax (tmax) | Day -1 until at least Day 7
Radioactivity in whole blood measured by Apparent Terminal Elimination Half-life (t1/2) | Day -1 until at least Day 7
Radioactivity in whole blood measured by Apparent total body clearance (CL/F) | Day -1 until at least Day 7
Radioactivity in whole blood measured by Apparent volume of distribution (Vz/F) | Day -1 until at least Day 7
Radioactivity in plasma measured by AUCinf | Day -1 until at least Day 7
Radioactivity in plasma measured by AUClast | Day -1 until at least Day 7
Radioactivity in plasma measured by Cmax | Day -1 until at least Day 7
Radioactivity in plasma measured by tmax | Day -1 until at least Day 7
Radioactivity in plasma measured by t1/2 | Day -1 until at least Day 7
Radioactivity in plasma measured by CL/F | Day -1 until at least Day 7
Radioactivity in plasma measured by Vz/F | Day -1 until at least Day 7
Radioactivity ratio of blood / plasma concentrations per time point and of Area under the plasma concentration (AUC) | Day -1 until at least Day 7
Excretion rate and cumulative excretion of radioactivity in urine | Day -1 until at least Day 7
Excretion rate and cumulative excretion of radioactivity in feces | Day -1 until at least Day 7
Total cumulative excretion of radioactivity in urine and feces | Day -1 until at least Day 7
ASP1707 in plasma measured by AUCinf | Day -1 until at least Day 7
ASP1707 in plasma measured by AUClast | Day -1 until at least Day 7
ASP1707 in plasma measured by Cmax | Day -1 until at least Day 7
ASP1707 in plasma measured by tmax | Day -1 until at least Day 7
ASP1707 in plasma measured by t1/2 | Day -1 until at least Day 7
ASP1707 in plasma measured by CL/F | Day -1 until at least Day 7
ASP1707 in plasma measured by Vz/F | Day -1 until at least Day 7
ASP1707 in urine measured by Amount excreted unchanged extrapolated to time = infinity (Aeinf) | Day -1 until at least Day 7
ASP1707 in urine measured by Amount excreted unchanged to last quantifiable sample (Aelast) | Day -1 until at least Day 7
ASP1707 in urine measured by Renal Clearance (CLR) | Day -1 until at least Day 7
ASP1707 in urine measured by Percentage of the dose excreted unchanged extrapolated to time = infinity (Aeinf%) | Day -1 until at least Day 7
ASP1707 in urine measured by Percentage of the dose excreted unchanged to last quantifiable sample (Aelast %) | Day -1 until at least Day 7

SECONDARY OUTCOMES:
Profiling of metabolites in plasma, urine and feces | Day -1 until at least Day 7
  This will be done separately from this study and will be reported in a separate report
Safety assessed by vital signs, 12-lead ECG, laboratory tests, adverse events, physical examination | Screening to ESV (up to Day 40)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Covance CRU Ltd., Leeds, United Kingdom